CLINICAL TRIAL: NCT02804100
Title: A Multi-centre Observational Study on Dynamic Changes of Circulating Tumor DNA in Late Stage NSCLC Patients Under Gefitinib Treatment
Brief Title: Dynamic Changes of Circulating Tumor DNA in Late Stage NSCLC Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Chunming Ding, Professor, Wenzhou Medical University
Other Study IDs: 4241616009G
Record Dates: First submitted 2016-06-14; First posted 2016-06-17 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Bronchial Neoplasms; Carcinoma, Bronchogenic; Lung Diseases; Lung Neoplasms
Keywords: Circulating Tumor DNA; Lung cancer; Plasma DNA
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Bronchial Neoplasms; Carcinoma, Bronchogenic; Lung Diseases; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A multi-centre observational, non-interventional study is to dynamically monitor the changes of circulating tumor DNA (ctDNA) in late stage NSCLC patients under Gefitinib treatment.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Histologically confirmed stage IIIB/IV NSCLC.
* Activating EGFR mutations (G719A/C/S; Exon 19 insertion/deletion; L858R; L861Q)
* Able to comply with the required protocol and followed-up procedures, and able to receive oral medications

Exclusion Criteria:

* Histologically confirmed small cell lung cancer or other metastatic tumors
* Patient had received prior chemotherapy or EGFR-TKIs treatment
* Patients who harbor Exon20 T790M mutation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NSCLC patients with activating EGFR mutations
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
dynamic changes of circulating tumor DNA in late stage NSCLC patients under Gefitinib treatment | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Wenfeng Li, Ph.D, Study Chair — First Affiliated Hospital of Wenzhou Medical University
Locations (1):
- Wenzhou Medical University, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yang Z, Li J, Hu Y, Chen M, Peng D, Zong D, Shang Q, Tao L, Zhao Y, Ni Y, Ye J, Xie Y, Yang L, Lin Q, Cai C, Xu N, Huang X, Dong X, Zhou Z, Yu Y, Shangguan Z, Xu Y, Ying W, Weng M, Yuan Z, Dong Z, Li J, Zheng Z, Pan J, Liu L, Ye J, Zhang Z, Li W, Zhu J, Jin S, Li Y, Ding C. Dynamics of Plasma EGFR T790M Mutation in Advanced NSCLC: A Multicenter Study. Target Oncol. 2019 Dec;14(6):719-728. doi: 10.1007/s11523-019-00682-0. PMID 31691892